CLINICAL TRIAL: NCT00485758
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled 36 Week Study to Evaluate the Efficacy and Safety of Extended Release (ER) Niacin/Laropiprant in Patients With Type 2 Diabetes
Brief Title: Extended Niacin/Laropiprant in Patients With Type 2 Diabetes (0524A-069)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-069; MK0524A-069; 2007_543
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Results first posted 2009-09-11 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — MK-0524; Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Other): Arm 1: One tablet of ER niacin/ laropiprant (1g) + one tablet of the run-in statin dose, advancing to ER niacin/laropiprant (2g) at Week 4 for the remainder of the study.
  Interventions: Drug: ER niacin/laropiprant
- 2 (Active Comparator): Arm 2: stable lipid-modifying regimen, adding Placebo ER niacin/laropiprant in week 4, for the duration of the study.
  Interventions: Drug: Comparator : placebo (unspecified)

INTERVENTIONS:
Drug: ER niacin/laropiprant — One tablet of ER niacin/laropiprant (1g); advancing to ER niacin/laropiprant (2g) at Week 4 for the remainder of the study 36 Weeks.
  Other Names: MK0524A; CORDAPTIVE™; laropiprant (+) niacin
  Arms: 1
Drug: Comparator : placebo (unspecified) — ER niacin/laropiprant Placebo
  Arms: 2

SUMMARY:
A study to assess the efficacy and tolerability of ER (Extended Release) niacin/laropiprant versus placebo in Type 2 Diabetes Mellitus patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 to 80 years with Type 2 Diabetes who are on a stable dose of antidiabetic medication for at least 3 months

Exclusion Criteria:

* Patients taking Cholestin, niacin (>50 mg/day), fibrate therapy, hormonal contraceptives, intermittent Hormone Replacement Therapy, or certain corticosteroids
* Patients with any of the following conditions: active liver disease or kidney disease, poorly controlled high blood pressure, active peptic ulcer, or other heart or blood diseases
* Patients with abnormal laboratory results from a blood test that will be given before starting the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 796 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] MacLean A, McKenney J, Scott R, Brinton E, Bays H, Mitchel Y, Paolini J, Giezek H, Vandormael K, Ruck RA, Gibson K, Sisk CM, Maccubbin D. Efficacy and safety of extended release niacin/laropiprant in patients with type 2 diabetes mellitus. Br J Cardiol. 2011;18(1):37-45.
- [Derived] Bays HE, Brinton EA, Triscari J, Chen E, Maccubbin D, MacLean AA, Gibson KL, Ruck RA, Johnson-Levonas AO, O'Neill EA, Mitchel YB. Extended-release niacin/laropiprant significantly improves lipid levels in type 2 diabetes mellitus irrespective of baseline glycemic control. Vasc Health Risk Manag. 2015 Feb 24;11:165-72. doi: 10.2147/VHRM.S70907. eCollection 2015. PMID 25750540
- [Derived] Bays HE, Shah A, Lin J, Sisk CM, Dong Q, Maccubbin D. Consistency of extended-release niacin/laropiprant effects on Lp(a), ApoB, non-HDL-C, Apo A1, and ApoB/ApoA1 ratio across patient subgroups. Am J Cardiovasc Drugs. 2012 Jun 1;12(3):197-206. doi: 10.2165/11631530-000000000-00000. PMID 22500948
- [Derived] Bays H, Giezek H, McKenney JM, O'Neill EA, Tershakovec AM. Extended-release niacin/laropiprant effects on lipoprotein subfractions in patients with type 2 diabetes mellitus. Metab Syndr Relat Disord. 2012 Aug;10(4):260-6. doi: 10.1089/met.2012.0005. Epub 2012 Mar 8. PMID 22400810
- [Derived] Bays H, Shah A, Dong Q, McCrary Sisk C, Maccubbin D. Extended-release niacin/laropiprant lipid-altering consistency across patient subgroups. Int J Clin Pract. 2011 Apr;65(4):436-45. doi: 10.1111/j.1742-1241.2010.02620.x. PMID 21401833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In:13-Aug-2007, Last Patient Last Visit:15-Jan-2009
  Ninety-four (94) sites participated: Australia 2 sites; Belgium 7 sites; Canada 6 sites; Ecuador 2 sites; Finland 2 sites; Germany 8 sites; Israel 4 sites; Italy 3 sites; Malaysia 5 sites; New Zealand 4 sites; Portugal 4 sites; Sweden 10 sites; Taiwan 5 sites; United States 32 sites
Pre-assignment Details: Patients with Type 2 Diabetes who were not at protocol specified low-density lipoprotein cholesterol goal of <115 milligrams/deciliter at screening, had a 4-week run-in period of lipid modifying therapy. In order to advance to randomization, patients had to meet the low-density lipoprotein cholesterol goal.
Groups:
- Extended Release Niacin/Laropiprant: One tablet of Extended Release Niacin/Laropiprant (1 gram/20 milligram) in addition to lipid modifying therapy. After 4 weeks, advanced to Extended Release Niacin/Laropiprant (2 gram/40 milligram).
  No adjustments were made to any lipid modifying regimen established during run-in until Week 12.
- Placebo: Matching placebo added to lipid modifying regimen and continued on this regimen for remainder of the study.
Period: Overall Study
Arm/Group | Extended Release Niacin/Laropiprant | Placebo
Started | 454 | 342
Completed | 298 | 277
Not Completed | 156 | 65
Not completed — Adverse Event | 102 | 31
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 5 | 1
Not completed — Physician Decision | 3 | 3
Not completed — Protocol Violation | 11 | 2
Not completed — Withdrawal by Subject | 32 | 27
Not completed — Study Terminated by Sponsor | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Release Niacin/Laropiprant | Placebo | Total
Number analyzed (Participants) | 454 | 342 | 796
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (9.3) | 62.0 (9.4) | 62.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 126 | 314
  Male | 266 | 216 | 482
Fasting Plasma Glucose [Mean (Standard Deviation); unit: milligrams/deciliter] | 132.0 (33.9) | 133.6 (32.4) | 132.7 (33.3)
High-density lipoprotein cholesterol [Mean (Standard Deviation); unit: milligrams/deciliter (mg/dl)] | 49.93 (13.49) | 50.26 (13.23) | 50.07 (13.37)
Low-density lipoprotein cholesterol [Mean (Standard Deviation); unit: milligrams/deciliter (mg/dl)] | 87.19 (20.54) | 85.22 (18.00) | 86.34 (19.50)
Triglycerides [Median (Full Range); unit: milligrams/deciliter (mg/dl)] | 126.00 [32.00 to 628.00] | 129.00 [39.00 to 509.00] | 127.00 [32.00 to 628.00]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change at Week (Wk) 12 Compared to Baseline (Bl) in Low-density Lipoprotein Cholesterol in Patients With Type 2 Diabetes When Compared to Placebo
Description: After 12 Weeks of treatment, to assess the reduction of low-density lipoprotein cholesterol in patients with Type 2 diabetes when compared to placebo
Time Frame: Baseline and 12 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change at Wk 12 compared to Bl
Arm/Group | Extended Release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 432 | 336
Percent change at Wk 12 compared to Bl | -15.8 [-18.4 to -13.2] | 2.1 [0.3 to 4.6]
Statistical Analysis 1: Comparison: Extended Release Niacin/Laropiprant vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Study times: 4, 8 and 12 weeks. Terms: treatment-by-time, gender-by-time and baseline low-density lipoprotein cholesterol -by-time interaction; Mean Difference (Final Values) = -17.9, 95% CI [-21.4 to -14.4], Standard Error of Mean 1.8

2. Secondary Outcome: Percent Change at Week (Wk) 12 Compared to Baseline (Bl) in High Density Lipoprotein Cholesterol in Patients With Type 2 Diabetes When Compared to Placebo
Description: After 12 weeks of treatment, to assess the increase of high-density lipoprotein cholesterol in patients with Type 2 diabetes when compared to placebo
Time Frame: Baseline and 12 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change at Wk 12 compared to Bl
Arm/Group | Extended Release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 432 | 336
Percent change at Wk 12 compared to Bl | 25.4 [23.4 to 27.5] | 2.2 [0.6 to 3.8]
Statistical Analysis 1: Comparison: Extended Release Niacin/Laropiprant vs Placebo; Test type: Superiority or Other; p < 0.001, Repeated Measures Analysis; Study times: 4, 8 and 12 weeks. Terms: treatment-by-time, gender-by-time and baseline high-density lipoprotein cholesterol -by-time interaction; Mean Difference (Final Values) = 23.2, 95% CI [20.7 to 25.7], Standard Error of Mean 1.3

3. Secondary Outcome: Percent Change at Week (Wk) 12 Compared to Baseline (Bl) in Triglycerides in Patients With Type 2 Diabetes When Compared to Placebo
Description: after 12 weeks of treatment, to assess the reduction of triglycerides in patients with Type 2 diabetes when compared to placebo
Time Frame: Baseline and 12 Weeks
Population: Full Analysis Set With at Least one Post-Titration Visit Measurement
Measure: Median (95% Confidence Interval); unit: Percent change at Wk 12 compared to Bl
Arm/Group | Extended Release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 400 | 328
Percent change at Wk 12 compared to Bl | -22.2 [-25.5 to -18.8] | 2.3 [-1.6 to 6.2]
Statistical Analysis 1: Comparison: Extended Release Niacin/Laropiprant vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Nonparametric Analysis of Covariance model based on Tukey's normalized ranks with term for treatment, gender and Tukey's normal score of baseline; Median Difference (Final Values) = -23.1, 95% CI [-27.2 to -18.9] — The median difference between treatments is based on the Hodges-Lehmann estimates of shift with a corresponding distribution-free Confidence Interval based on Wilcoxon's rank

ADVERSE EVENTS:
Description: 7 randomized patients took no study drug dose and were not included in the safety follow-up
Arm/Group | Extended Release Niacin/Laropiprant | Placebo
Serious Adverse Events (participants affected / at risk) | 26/449 | 24/340
Other Adverse Events (participants affected / at risk) | 251/449 | 113/340
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Extended Release Niacin/Laropiprant (N=449) | Placebo (N=340)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 2
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 2 | 0
Cataract (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Extended Release Niacin/Laropiprant (N=449) | Placebo (N=340)
Diarrhoea (Gastrointestinal disorders) | 41 | 21
Nausea (Gastrointestinal disorders) | 24 | 12
Nasopharyngitis (Infections and infestations) | 33 | 25
Upper respiratory tract infection (Infections and infestations) | 28 | 24
Blood glucose increased (Investigations) | 52 | 14
Headache (Nervous system disorders) | 20 | 18
Pruritus (Skin and subcutaneous tissue disorders) | 71 | 9
Rash (Skin and subcutaneous tissue disorders) | 26 | 5
Flushing (Vascular disorders) | 79 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.